CLINICAL TRIAL: NCT01983618
Title: Impact of Interscalene Nerve Block on Cerebral Perfusion During Surgery in the Beachchair Position Under General Anesthesia
Brief Title: Impact of Interscalene Nerve Block on Cerebral Perfusion During Surgery in the Beachchair Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13.226
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Cerebral Ischemia
Keywords: Cerebral ischemia; Beachchair position; Interscalene nerve block
MeSH Terms: conditions — Brain Ischemia | interventions — Catheters

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interscalene catheter (Placebo Comparator): No block will be performed prior to surgery. An interscalene catheter will be inserted under ultrasound guidance by the anesthesiologist before the induction of anesthesia. Local anesthetics will only be administered once all TCD assessments are completed but prior to the end of surgery.
  Interventions: Procedure: Interscalene catheter
- Interscalene nerve block and catheter (Experimental): The anesthesiologist will perform the interscalene nerve block and insert an interscalene catheter under ultrasound guidance before induction of anesthesia. A standardized mixture of bupivacaine, lidocaine and epinephrine will be administered prior to surgery.
  Interventions: Procedure: Interscalene nerve block and catheter

INTERVENTIONS:
Procedure: Interscalene nerve block and catheter
  Arms: Interscalene nerve block and catheter
Procedure: Interscalene catheter
  Arms: Interscalene catheter

SUMMARY:
Beachchair position is used by many orthopaedic surgeons for shoulder surgery. Most patients undergoing surgery in this position have no complications. However, reported cases of postoperative neurological deficits have highlighted the risk of cerebral and spinal cord ischemia. The etiology of such complications remains unclear. The most plausible explanation for these events would be intraoperative hypotension followed by cerebral hypoperfusion.

General anesthesia is commonly used for shoulder surgery in conjunction with interscalene brachial plexus blockade. During the block, local anesthetic's spread is frequently observed leading to a block of sympathetic fibres. Since all nerves located in the head and neck area go through the stellate ganglion, its block will cause a sympathetic denervation and a decrease of the peripheral vascular resistance, thus increasing the circulation in cerebral blood vessels. In normal situations, there is a vasoconstriction of the cerebral blood vessels in response to a sympathetic stimulation and a vasodilation if sympathetic fibres are blocked.

Transcranial Doppler (TCD) is a non-invasive examination that provides a reliable evaluation of intracranial blood flow in real-time. It can help to detect sudden changes in perfusion and identify potential embolic events. Some studies using TCD have shown an increased ipsilateral cerebral blood flow (CBF) secondary to a reduced vascular tone associated with a stellate ganglion block. Others have shown a reduction of contralateral CBF that could theoretically increase the risk of ischemia in the affected area.

This study will assess the role of interscalene nerve blockade in the protection of cerebral ischemia and preservation of cerebral autoregulation. This study will also aim to identify changes in contralateral CBF.

The investigators hypothesize that:

1. Interscalene nerve block will increase CBF
2. Interscalene nerve block will not decrease contralateral CBF
3. Cerebral autoregulation will be preserved under general anesthesia in conjunction with an interscalene nerve block in this setting.

DETAILED DESCRIPTION:
Prior to surgery, each patient will undergo a baseline bilateral TCD examination in supine position. If the Doppler's results are satisfactory, the patient will then be randomized and proceed to the next step. In case of inadequate results, the patient's participation to the study will be terminated.

The interscalene nerve block and the insertion of the interscalene catheter will be performed according to randomization. In the interscalene nerve block and catheter group, the attending anaesthesiologist will assess the success of the block and record the presence or absence of Horner's syndrome. The transcranial Doppler operator will be blinded to these observations. Following the insertion of the interscalene catheter, the patient will undergo a second bilateral TCD in supine position before induction of anesthesia.

The anesthetic technique and monitoring will be standardized. After the induction of anesthesia, a bilateral TCD will be performed with the patient in supine position. Another examination will be performed under general anesthesia immediately after and 30 minutes following the installation of the patient in the beachchair position. A last TCD will be performed after a reduction of end-tidal carbon dioxide at 30 mm Hg.

For each examination, the arterial blood pressure must be stabilized for at least 5 minutes before the Doppler can be initiated. Arterial blood pressure will be measured during each examination. Type, duration of surgery and beachchair position will be recorded. Vasopressor therapy will be noted. Body temperature, end-tidal carbon dioxide and minimum alveolar concentration of desflurane will be collected during each examination performed under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for shoulder surgery in the sitting position
* Surgery of the shoulder and clavicular area, eligible to an interscalene nerve block
* American Society of Anesthesiologists (ASA) physical status 1-3

Exclusion Criteria:

* Carotid artery stenosis
* History of stroke or other significant central nervous system lesion
* Inadequate temporal window to perform transcranial Doppler
* Contraindication to interscalene nerve block
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow in the median cerebral artery | From arrival in the operating theatre until the end of surgery. Patients will be followed for an average of 3 hours.
  Cerebral blood flow will be assessed using the transcranial Doppler. Because the bones of the skull block the transmission of ultrasound, region with thinner walls must be used for analyzing. For this reason, recording will be performed in the temporal region above the zygomatic arch.

SECONDARY OUTCOMES:
Arterial blood pressure | From arrival in the operating theatre until the end of surgery. Patients will be followed for an average of 3 hours.
  Arterial blood pressure will be measured during each TCD.
Body temperature | From induction of anesthesia until the end of surgery. Patients will be followed for an average of 2 hours.
  Body temperature will be recorded at every TCD performed following induction of general anesthesia.
End-tidal carbon dioxide | From induction of anesthesia until the end of surgery. Patients will be followed for an average of 2 hours.
  End-tidal carbon dioxide will be recorded at every TCD performed following induction of general anesthesia.
Minimum alveolar concentration (MAC) of Desflurane | From induction of anesthesia until the end of surgery. Patients will be followed for an average of 2 hours.
  Minimum alveolar concentration of Desflurane will be recorded at every TCD performed following induction of general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Garneau, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada